CLINICAL TRIAL: NCT01388283
Title: Inflammatory Markers in Pregnant Women Destined to Develop Preeclampsia
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Oslo University Hospital, Department of Medical Biochemistry
Other Study IDs: INMARPE11
Record Dates: First submitted 2011-06-30; First posted 2011-07-06 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-06

CONDITIONS: Preeclampsia
Keywords: prognostic marker
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the predictive role of serum inflammatory markers in pregnant women who subsequently develop preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* caucasian,
* nulliparous

Exclusion Criteria:

* preexisting cardiovascular diseases,
* diabetes,
* hypertension,
* inflammatory bowel diseases,
* serious organ diseases, and
* development of separate gestational diabetes and/or hypertension.

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Case-control study consisting of 43 women developping preeclampsia and 86 women not developping this disorder. All were of Caucasian origin and were nulliparous.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 1999-01; Primary Completion 2004-05 (Actual); Study Completion 2011-06 (Actual)